CLINICAL TRIAL: NCT00057421
Title: Impact of Tuberculosis on HIV Infection in Uganda
Brief Title: Tuberculosis in HIV Infected Patients in Uganda
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AI032414 (NIH); R01AI032414 (NIH)
Record Dates: First submitted 2003-04-01; First posted 2003-04-03 (Estimated); Last update posted 2007-09-18 (Estimated); Status verified 2007-08

CONDITIONS: Tuberculosis; HIV Infections
Keywords: Tuberculosis; HIV infection; Prednisolone; Safety; Immune activation
MeSH Terms: conditions — Tuberculosis; HIV Infections | interventions — Prednisolone

INTERVENTIONS:
Drug: prednisolone

SUMMARY:
This was a clinical trial in HIV infected patients with tuberculosis. The study assessed whether the addition of prednisolone, a type of steroid medication, to the standard treatment for tuberculosis improved immune and viral outcomes in the patients. The study demonstrated that prednisolone increased the CD4 cell count as was hoped, but the beneficial effect was short-lived and was gone within 4 months of stopping therapy. Therefore, the use of prednisolone for tuberculosis in HIV infected patients is not recommended at this time.

DETAILED DESCRIPTION:
Recent observations from retrospective cohort studies indicate that HIV-associated tuberculosis (TB) is associated with reduced survival and increased rate of opportunistic infections compared to CD4-matched controls. Mounting evidence from immunologic and virologic studies supports the concept of co-pathogenesis, in which cytokines such as tumor necrosis factor alpha (TNF alpha) are over-expressed during the course of TB and stimulate viral replication in latently infected cells, possibly leading to greater viral load.

Glucocorticoids are potent inhibitors of cytokines, including TNF, and clinicians have extensive experiences with their use in HIV infection. Although corticosteroid use in HIV infection has a record of safety, the safety and bioavailability of corticosteroids in HIV/TB coinfection has not been established.

This study evaluated the change in viral load and CD4 count in HIV infected patients with TB who were treated with oral prednisolone. The study found that the viral load increased slightly when prednisolone was administered and that patients receiving prednisolone cleared their tuberculosis more rapidly. Although there was some benefit to using prednisolone in these patients, the benefit was short-lived and was gone within 4 months of stopping therapy.

ELIGIBILITY:
Inclusion Criteria

* Pulmonary TB (smear positive)
* HIV infected
* Residence within 20 km of Kampala city
* Allows frequent blood specimens to be drawn

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 190
Dates: Start 1998-11; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Whalen, Principal Investigator — Case Western Reserve University
Locations (1):
- Mulago Hospital Tuberculosis Clinic, Kampala, Uganda